CLINICAL TRIAL: NCT00262145
Title: Ability of a Tea Leaf Extracts Preparation to Slow Down Carbohydrate and Fat Uptake in Human
Brief Title: Ability of a Tea Leaf Extracts Preparation to Slow Down Carbohydrate and Fat Absorption
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NatureGen (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NA051001
Record Dates: First submitted 2005-12-05; First posted 2005-12-06 (Estimated); Last update posted 2005-12-06 (Estimated); Status verified 2005-10

CONDITIONS: Diabetes; Overweight
Keywords: glucose; lipid; diabetes; overweight
MeSH Terms: conditions — Diabetes Mellitus; Overweight

INTERVENTIONS:
Drug: tea extracts

SUMMARY:
Objective - A variety of herbal, over-the-counter preparations of tea leaves are said to reduce the rate of absorption of fat ( allegedly via inhibition of pancreatic lipase) and carbohydrate (via inhibition of carbohydrate digestion and blocking of glucose transport by the intestinal mucosa). There has been some study of the ability of these products to reduce the blood glucose increase observed after a carbohydrate meal and to reduce blood cholesterol levels in chronic studies. The purpose of the present study is to objectively determine if one cup of "tea" made from a combination of three types of tea leaves (mulberry, black and green tea) can cause malabsorption of carbohydrate and fat taken in conjunction with the tea.

Research Design - The study will consist of a double blind, placebo controlled crossover study in 20 healthy subjects. On one of two days (one week apart) the subjects will ingest a standard meal consisting of 30 g of sucrose (in the tea) and 30 g of starch in the form of white rice plus 10 g of fat as butter. To measure triglyceride absorption, each meal will also contain 250 mg of 13-C labeled triolein. Triolein is a commonly ingested fat consisting of glycerol bound to three oleic acids. 13-C is a stable (non-radioactive) isotope of carbon. On one of the test days the subjects (randomly) will concurrently consume the active preparation, a tea containing extracts of the three types of tea leave described above plus the meal, and on the other test day they will consume the meal with a liquid placebo preparation (warm water, sugar and food coloring). Subjects will provide a breath sample before and at hourly intervals for 8 hours after ingestion of the meal. Carbohydrate malabsorption will be determined by the hydrogen concentration in the breath samples and fat malabsorption by the concentration of 13-CO2 in the breath samples.

Clinical Significance - An increase in breath hydrogen indicates carbohydrate malabsoption and a low 13-CO2 indicates lipid malabsorption. Objective evidence that the tea leaf extract actually induces carbohydrate and/or fat malabsorption could provide the basis for further studies.

DETAILED DESCRIPTION:
One of the commonly cited beneficial effects of tea is its ability to induce weight loss. Support for this contention include a controlled human trial showing increased weight loss when tea was added to a dietary regimen, and a mouse study demonstrating that administration of a tea extract with a high fat diet eliminated the weight gain observed in the absence of tea. Several different mechanisms have been postulated to account for this weight control. Multiple studies have reported modest increases in energy expenditure associated with ingestion of oolong or green teas. In addition, tea could inhibit the absorption of carbohydrate and/or fat. Studies supporting the possibility of carbohydrate malabsorption include a in vitro studies showing that constituents of tea inhibit the activity of carbohydrate digesting enzymes (α-amylase and α-glucosidase, and the mucosal uptake of glucose via an interaction with sodium dependent glucose transporters. The in vitro demonstration that tea extracts inhibit pancreatic lipase activity suggests that tea might interfere with triglyceride absorption.

However, there have been no in vivo studies in humans or animals showing that tea preparations actually are capable of causing malabsorption of either carbohydrate or fat. In the present study, we utilized measurements of breath H2 and 13CO2 to investigate the ability of a mixture of black, green and mulberry tea leaf extracts to induce malabsorption of carbohydrate and fat in healthy volunteers.

Protocol - The study group consisted of 20 healthy volunteers (ages 23 to 52, 10 females and 10 males). The subjects fasted after their usual dinner on the day preceding the study until the following morning (approximately 8 am) when the experiments were performed. After collection of baseline breath samples for H2 and 13CO2 analysis, the subjects ingested the test meal that consisted of cooked white rice and butter. The rice was boiled for20 minutes, and then individual portions (176 g, which contained 50 g of carbohydrate) were weighed and frozen with 10g of butter. Immediately prior to ingestion, the meals were warmed in a microwave oven, and 0.2 g of 1,1,1-13C-triolein (Cambridge Isotope Laboratories, Andover, MA) was thoroughly mixed into the meal. Concurrent with ingestion of the meal, the subjects randomly were assigned to drink either 500 ml of the warm active tea preparation containing 10 g of sucrose or 500 ml of a placebo preparation that also contained 10 g of sucrose. Breath samples were then collected at hourly intervals for eight hours. At the end of each test period, subjects were asked to rate a variety of symptoms including nausea, bloating, abdominal discomfort, and rectal gas (as well as obfuscating symptoms) on a previously described linear scale that ranged from zero (none) to 4 (severe). In addition, the number of loose bowel movements were noted. One week later the test was repeated with the subjects receiving the opposite preparation from that used in the initial study. The study was approved by the Human Studies Subcommittee of the Mpls. VA Medical center and informed consent was obtained from all subjects.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 60 years old, healthy individuals

Exclusion Criteria:

* pregnant women

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20
Dates: Start 2005-10; Study Completion 2005-11

PRIMARY OUTCOMES:
glucose and lipid uptake

SECONDARY OUTCOMES:
lipid metabolism

CONTACTS AND LOCATIONS:
Overall Officials: Michael D Levitt, M.D., Principal Investigator — VA Medical Center, Minneapolis, MN
Locations (1):
- VA Medical Center, Minneapolis, Minnesota, United States